CLINICAL TRIAL: NCT03347942
Title: Clinical Study Randomized of the Effects of the Administered Time of Meal on the Treatment of Overweight and Obesity
Brief Title: Effects of the Administered Time of Meal on the Treatment of Overweight and Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0327
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-09

CONDITIONS: Feeding Behavior; Diet, Reducing; Eating
Keywords: Overweight; Obesity; Satiety; Cardiovascular risk
MeSH Terms: conditions — Feeding Behavior; Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized and controlled clinical trial in adults of both sexes, overweight and obese who accepted to participate in the research at the Hospital de Clínicas in the city of Porto Alegre. Individuals will be divided into two paired groups for age, gender and waist diameter. These two groups will be randomized by lottery.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded, as they will be instructed to perform the intervention in the control of meal time. This is a limitation of the study design, however, it is expected to minimize the bias by not explaining to the participants what is expected by the intervention of the research. The researcher, who will measure the outcomes, will not know to which group the individual belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): During a period of 30 days the research participant in the intervention group will be instructed to wait at least 20 minutes after finishing the first portion of meals previously considered sufficient by the individual before being served again if he or she feels the need.
  Interventions: Behavioral: Intervention group
- Control (Other): The control group will also serve the dish the same way, but you can serve additional portion without waiting.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Intervention group — Wait at least 20 minutes after finishing the first portion of meals previously considered sufficient by the individual before serving again if he or she feels the need. The intervention time will be monitored by the participants themselves, who will be instructed by the researcher when the methodology to be performed.
  Arms: Intervention
Other: Control group — The control group will also serve the dish of the form, but can serve additional portion without waiting.
  Arms: Control

SUMMARY:
Objectives: To evaluate the impact of the meal time administered on the body weight of adult individuals of both sexes, being overweight and obese.

Experimental design: randomized controlled trial. Place of research: Hospital de Clínicas de Porto Alegre, Porto Alegre, RS, Brazil.

Materials and methods: Anthropometric data, blood pressure, waist diameter will be measured; venous blood samples will be collected and stored for glucose, total cholesterol, triglycerides, HDL-cholesterol, urea, creatinine and ALT in serum.

Intervention: Wait at least 20 minutes after finishing the first portion of meals, previously considered sufficient by the individual before serving again. The control group will also serve the dish the same way, but you can serve additional portion without waiting.

Measurements: P values less than 0.05 will be considered statistically significant.

Expected results: Weight loss, decrease in anthropometric markers and risk factors for cardiovascular diseases.

DETAILED DESCRIPTION:
Introduction: The increasing rates of overweight and obesity in the world population have worried health professionals about their quality and life expectancy. Intervention methods such as weight management programs can promote eating behaviors more suited to the energy needs of these individuals.

Objectives: To evaluate the impact of the meal time administered on the body weight of adult individuals of both sexes, overweight and obese.

Experimental design: randomized controlled trial. Place of research: Hospital de Clínicas de Porto Alegre, Porto Alegre, RS, Brazil.

Participants: Adults of both sexes. Materials and methods: Individuals will be invited to participate and will receive a free and informed consent form. If they agree, anthropometric data, blood pressure, waist diameter will be measured; venous blood samples will be collected and stored for glucose, total cholesterol, triglycerides, HDL-cholesterol, urea, creatinine and ALT in serum.

Intervention: Wait at least 20 minutes after finishing the first portion of meals, previously considered sufficient by the individual before serving again. The control group will also serve the dish the same way, but you can serve additional portion without waiting.

Measurements: The Kolmogorov-Smirnoff tests will be used to evaluate the distribution of continuous variables, and Student's t test, Mann-Whitney, and chi-square test, when appropriate. Values of p less than 0.05 will be considered statistically significant.

Expected results: Adults randomized to receive the intervention will gain weight loss, decrease in anthropometric markers and risk factors for cardiovascular diseases.

Project cost / benefit: Low cost and risk study that will contribute to the development of actions and programs related to the reduction of risk factors due to overweight and disease prevention.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obesity grade I, according to WHO criteria (1998).

Exclusion Criteria:

* Normal weight, obesity> grade I;
* Use of appetite-enhancing medications such as glucocorticoids, tricyclic antidepressants, antipsychotics, mood modulators and anticonvulsants, or reduce body weight , such as anorexigenics, and antidiabetics that can modify body weight;
* In follow-up or nutritional intervention already established and;
* Refusal to sign the informed consent form.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Mean body weight | 30 days
  * Measurement of body weight in kilograms - will be carried out on the balance of Toledo® brand with a capacity of 200 kg, after urinating.
  * The individual will keep his body erect, with arms hanging over the body and heels attached.
  * Participants should only be in their underwear and disposable surgical dress, barefoot.

SECONDARY OUTCOMES:
Cardiovascular risk assessment scores | 30 days
  The calculation will be done with the CV Risk Calculator tool of the American College of Cardiology and the American Cardiology Association to obtain the percentage (%) risk for acute myocardial infarction or stroke in ten years.
Waist diameter values | 30 days
  * It will be obtained with flexible tape and inelastic (in centimeters), with the individual standing erect, arms extended along the body and feet together.
  * The tape will be positioned at the midpoint between the iliac crest and the outer side of the last rib.

CONTACTS AND LOCATIONS:
Overall Officials: Tania W Furlanetto, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No